CLINICAL TRIAL: NCT07040657
Title: Comparison of Two-Point and Four-Point Cervical Injection Techniques Using Methylene Blue for Sentinel Lymph Node Mapping in Endometrial Cancer
Brief Title: Comparison of Two-Position and Four-Position Cervical Injection Techniques for Sentinel Lymph Node Mapping in Endometrial Cancer Using Methylene Blue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, İbrahim Yalçın, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 693-SBKAEK
Record Dates: First submitted 2025-06-05; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Endometrial Neoplasms; Endometrial Cancer Stage I; Sentinel Lymph Node; Metastasis
Keywords: endometrial neoplasm; methylene blue; metastasis; cervix
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
Who Masked: Participant, Care Provider
Masking Description: To minimize bias and ensure the reliability of study results, both participants and care providers will be blinded to group allocation. The surgeon administering the injection and the pathologist evaluating lymph node samples will not be informed whether the participant received the two-point or four-point cervical injection. This double-masking approach enhances the objectivity of care delivery and outcome assessment, thereby strengthening the validity of the findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2- Point Methylene Blue Injection (Experimental): In the 2-point injection arm, participants will receive the standard sentinel lymph node (SLN) mapping technique using methylene blue. The procedure involves injecting methylene blue dye into two specific locations on the cervix:
  At the 3 o'clock position At the 9 o'clock position
  Interventions: Procedure: Sentinel Lymph Node Detection/Cervical Methylene Blue Injection
- 4- Point Methylene Blue Injection (Active Comparator): In the 4-point injection arm, participants will receive the standard sentinel lymph node (SLN) mapping technique using methylene blue. The procedure involves injecting methylene blue dye into two specific locations on the cervix:
  At the 2 o'clock position At the 4 o'clock position At the 8 o'clock position At the 10 o'clock position
  Interventions: Procedure: Sentinel Lymph Node Detection/Cervical Methylene Blue Injection

INTERVENTIONS:
Procedure: Sentinel Lymph Node Detection/Cervical Methylene Blue Injection — Sentinel Lymph Node (SLN) detection using cervical methylene blue injection is a surgical technique designed to identify the primary lymph nodes responsible for draining the uterus in patients with endometrial cancer. The procedure involves injecting methylene blue dye into specific locations within the cervical stroma to enable lymphatic uptake. The dye subsequently travels through the lymphatic channels, allowing for intraoperative visual identification of the sentinel nodes. This targeted approach facilitates selective SLN excision for pathological evaluation, providing critical information about lymphatic involvement while minimizing the extent of surgical dissection. The effectiveness of SLN mapping is contingent upon the accuracy of the injection technique and the anatomical distribution of lymphatic drainage.

SUMMARY:
This clinical trial evaluates lymph node mapping in newly diagnosed endometrial cancer patients undergoing surgery. The standard technique uses a 2-point methylene blue cervical injection. The study aims to determine if increasing injection points improves mapping success.

DETAILED DESCRIPTION:
In recent years, Sentinel Lymph Node (SLN) mapping has become a key focus in improving surgical outcomes for endometrial cancer. While methylene blue is a cost-effective option for SLN mapping, its detection rates remain suboptimal. This study aims to evaluate whether increasing the injection points from the standard 2-point to a 4-point methylene blue injection improves SLN mapping success.

This randomized controlled trial will include patients with preoperative stage I endometrial carcinoma. Participants will be randomized into two groups: one group will receive a 2-point methylene blue cervical injection, and the other group will receive a 4-point injection.

The primary endpoint is the difference in SLN detection rates between the two techniques. Findings from this study will provide detailed insights into whether the 4-point injection offers a significant advantage over the standard 2-point method.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with stage I endometrial cancer based on CT and PET-CT imaging.
* Individuals with a pathologically confirmed diagnosis of stage I endometrial cancer.

Exclusion Criteria:

Medical Conditions

* Individuals diagnosed with dementia.
* Individuals with allergies to methylene blue or iodine.
* Individuals who have received active treatment for another malignancy within the past five years.
* Inability to successfully perform PLD (pelvic lymphadenectomy) or history of prior PLD.
* Women with multiple and confluent lymph nodes identified as positive on FDG-PET/CT (such cases are not considered stage I).

Cancer-Related Conditions

* Individuals with clinically or radiologically identified positive lymph nodes or metastatic disease.
* Individuals with a history of pelvic dissection and/or radiation therapy.
* Individuals with advanced cervical or uterine cancer.
* Individuals with T3/T4 lesions.
* Individuals with cervical tumors larger than 2 cm.

Organ Dysfunction

• Individuals with hepatic dysfunction and a MELD score ≥ 10 and creatinine ≥ 2·0 mg/dl patients.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is limited to female participants, as it focuses on sentinel lymph node (SLN) mapping in patients with endometrial cancer, a disease that exclusively affects individuals with a uterus. Male participants are not eligible for inclusion in this study.
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Sentinel Lymph Node (SLN) Detection Rate | 1 day
  The detection rate will be measured as the number of sentinel lymph nodes identified using methylene blue divided by the total number of lymph nodes excised during surgery. Comparison will be made between the two-point and four-point cervical injection techniques. (Unit of Measure: Proportion (%))
Sensitivity of SLN Biopsy for Detecting Lymph Node Metastases | 1 day
  Sensitivity will be calculated as the proportion of true positive SLNs (confirmed by histopathology) over the total number of lymph nodes with metastases.
  (Unit of Measure: Percentage (%))
Specificity of SLN Biopsy for Detecting Lymph Node Metastases | 1 day
  Description: Specificity will be calculated as the proportion of true negative SLNs over all lymph nodes without metastasis.
  (Unit of Measure: Percentage (%))
Rate of Positive SLNs Detected | 1 day
  Proportion of SLNs identified as positive for metastasis in each injection technique group. (Unit of Measure: Proportion (%))

SECONDARY OUTCOMES:
Procedure Duration | 1 day
  Total time in minutes from injection to identification of sentinel lymph nodes (SLNs), recorded and compared between two-point and four-point cervical injection techniques. (Unit of Measure: Minutes)
Complications and Side Effects - Injection-Related Side Effects | 1 month
  Incidence of side effects related to methylene blue injection (e.g., allergic reaction, local pain, or discoloration at the injection site), recorded during and after the procedure. (Unit of Measure: Number of events and proportion (%))
SLN Anatomical Distribution | 1 day
  Number and proportion of detected SLNs located in specific anatomical regions (e.g., pelvic, para-aortic) for each injection technique. (Unit of Measure: Number and Proportion (%))
Surgical Complications | 1 month
  Incidence of postoperative complications related to SLN mapping, including infection, hematoma, and lymphedema. (Unit of Measure: Number of events and proportion (%))

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University, Ankara
  - Dokuz Eylul University, Izmir

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD related to the primary and secondary outcomes will be shared upon reasonable request. Access will be granted for academic and scientific research purposes, subject to approval by the study investigators and compliance with ethical and regulatory guidelines. A data-sharing agreement will be required to ensure proper use and confidentiality of the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Sehnal B, Waldauf P, Matej R, Hruda M, Robova H, Drozenova J, Pichlik T, Zapletal J, Rob L, Halaska MJ. Comparison of tracer application methods for sentinel lymph node detection in open surgery patients with endometrial cancer: a retrospective cohort study. BMC Cancer. 2025 Apr 8;25(1):638. doi: 10.1186/s12885-025-14037-8. PMID 40200256
- [Background] Holloway RW, Abu-Rustum NR, Backes FJ, Boggess JF, Gotlieb WH, Jeffrey Lowery W, Rossi EC, Tanner EJ, Wolsky RJ. Sentinel lymph node mapping and staging in endometrial cancer: A Society of Gynecologic Oncology literature review with consensus recommendations. Gynecol Oncol. 2017 Aug;146(2):405-415. doi: 10.1016/j.ygyno.2017.05.027. Epub 2017 May 28. PMID 28566221
- [Background] Salman L, Cusimano MC, Marchocki Z, Ferguson SE. Sentinel lymph node mapping in endometrial cancer: Current evidence and practice. J Surg Oncol. 2024 Jan;129(1):117-119. doi: 10.1002/jso.27550. Epub 2023 Dec 7. PMID 38059317
- [Background] Leitao MM Jr, Zhou QC, Gomez-Hidalgo NR, Iasonos A, Baser R, Mezzancello M, Chang K, Ward J, Chi DS, Long Roche K, Sonoda Y, Brown CL, Mueller JJ, Gardner GJ, Jewell EL, Broach V, Zivanovic O, Dowdy SC, Mariani A, Abu-Rustum NR. Patient-reported outcomes after surgery for endometrial carcinoma: Prevalence of lower-extremity lymphedema after sentinel lymph node mapping versus lymphadenectomy. Gynecol Oncol. 2020 Jan;156(1):147-153. doi: 10.1016/j.ygyno.2019.11.003. Epub 2019 Nov 25. PMID 31780238
- [Background] Terada S, Tanaka T, Murakami H, Tsuchihashi H, Toji A, Daimon A, Miyamoto S, Nishie R, Ueda S, Hashida S, Morita N, Maruoka H, Konishi H, Kogata Y, Taniguchi K, Komura K, Ohmichi M. Lymphatic Complications Following Sentinel Node Biopsy or Pelvic Lymphadenectomy for Endometrial Cancer. J Clin Med. 2023 Jul 7;12(13):4540. doi: 10.3390/jcm12134540. PMID 37445574
- [Background] Altin D, Taskin S, Ortac F, Tokgozoglu N, Vatansever D, Guler AH, Gungor M, Tasci T, Bese T, Turan H, Kahramanoglu I, Yalcin I, Celik C, Demirkiran F, Kose F, Arvas M, Ayhan A, Taskiran C. Diagnostic accuracy of sentinel node biopsy in non-endometrioid, high-grade and/or deep myoinvasive endometrial cancer: A Turkish gynecologic oncology group study (TRSGO-SLN-006). Gynecol Oncol. 2022 Mar;164(3):492-497. doi: 10.1016/j.ygyno.2022.01.009. Epub 2022 Jan 13. PMID 35033380
- [Background] Niikura H, Kaiho-Sakuma M, Tokunaga H, Toyoshima M, Utsunomiya H, Nagase S, Takano T, Watanabe M, Ito K, Yaegashi N. Tracer injection sites and combinations for sentinel lymph node detection in patients with endometrial cancer. Gynecol Oncol. 2013 Nov;131(2):299-303. doi: 10.1016/j.ygyno.2013.08.018. Epub 2013 Aug 27. PMID 23988415
- [Background] Geppert B, Lonnerfors C, Bollino M, Arechvo A, Persson J. A study on uterine lymphatic anatomy for standardization of pelvic sentinel lymph node detection in endometrial cancer. Gynecol Oncol. 2017 May;145(2):256-261. doi: 10.1016/j.ygyno.2017.02.018. Epub 2017 Feb 10. PMID 28196672
- [Background] Perrone AM, Casadio P, Formelli G, Levorato M, Ghi T, Costa S, Meriggiola MC, Pelusi G. Cervical and hysteroscopic injection for identification of sentinel lymph node in endometrial cancer. Gynecol Oncol. 2008 Oct;111(1):62-7. doi: 10.1016/j.ygyno.2008.05.032. Epub 2008 Jul 14. PMID 18625518
- [Background] Dick A, Perri T, Kogan L, Brandt B, Meyer R, Levin G. Sentinel lymph node mapping in endometrial cancer: A comparison of main national and international guidelines. Int J Gynaecol Obstet. 2023 Jan;160(1):220-225. doi: 10.1002/ijgo.14307. Epub 2022 Jul 5. PMID 35700068
- [Background] Fotopoulou C, Ind T, Baldwin P, Crawford R, Devaja O, Dobbs S, Frost J, Gajjar K, Ganesan R, Kaushik S, Morrison J, Nobbenhuis M, Ratnavelu N, Rolland P, Singh N, Taylor A, Sundar S, Nordin A. Sentinel lymph node consensus document of the British Gynaecological Cancer Society for endometrial, vulvar, and cervical cancers. Int J Gynecol Cancer. 2019 Nov;29(9):1348-1350. doi: 10.1136/ijgc-2019-000798. No abstract available. PMID 31685556
- [Background] Dioun S, Chen L, Melamed A, Gockley A, St Clair CM, Hou JY, Khoury-Collado F, Hershman DL, Wright JD. Uptake and outcomes of sentinel lymph node mapping in women undergoing minimally invasive surgery for endometrial cancer. BJOG. 2022 Aug;129(9):1591-1599. doi: 10.1111/1471-0528.17085. Epub 2022 Jan 25. PMID 34962708
- [Background] Baiocchi G, Andrade CEMC, Ribeiro R, Moretti-Marques R, Tsunoda AT, Alvarenga-Bezerra V, Lopes A, Costa RLR, Kumagai LY, Badiglian-Filho L, Faloppa CC, Mantoan H, De Brot L, Dos Reis R, Goncalves BT. Sentinel lymph node mapping versus sentinel lymph node mapping with systematic lymphadenectomy in endometrial cancer: an open-label, non-inferiority, randomized trial (ALICE trial). Int J Gynecol Cancer. 2022 May 3;32(5):676-679. doi: 10.1136/ijgc-2022-003378. PMID 35236752
- [Background] Sozzi G, Fanfani F, Berretta R, Capozzi VA, Uccella S, Buono N, Giallombardo V, Di Donna MC, Monterossi G, Restaino S, Capasso I, Dinoi G, Scambia G, Chiantera V. Laparoscopic sentinel node mapping with intracervical indocyanine green injection for endometrial cancer: the SENTIFAIL study - a multicentric analysis of predictors of failed mapping. Int J Gynecol Cancer. 2020 Nov;30(11):1713-1718. doi: 10.1136/ijgc-2020-001724. Epub 2020 Aug 31. PMID 32868384